CLINICAL TRIAL: NCT06450444
Title: Randomized, Double-blind, Sham-controlled Trial to Investigate Combined Occipital and Supra-orbital Neuromodulation in Resistant Migraine. The RECLAIM Study.
Brief Title: The RECLAIM Study.
Acronym: RECLAIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salvia BioElectronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCI-03-RM
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Migraine; High Frequency Episodic Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Active Stimulation
  Interventions: Device: PRIMUS
- Control Group (Other): Sham stimulation
  Interventions: Device: PRIMUS

INTERVENTIONS:
Device: PRIMUS — The Salvia PRIMUS System is designed to provide subcutaneous neurostimulation to the branches of the trigeminal and occipital nerves.

SUMMARY:
The purpose of this study is to evaluate the safety and performance, including clinical benefit, of the PRIMUS System for the treatment of Resistant Migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine as defined by the ICHD-3 Classification (with or without aura) with a history of chronic or high-frequency episodic migraine for at least 1 year prior to screening
* Failure of 3 or more preventive pharmacological therapies
* Stable on preventive migraine treatments
* Psychologically stable

Exclusion Criteria:

* Concomitant invasive or non-invasive neuromodulation
* Previous exposure to an implantable neuromodulation device for headache
* Have an existing active implantable medical device nearby the implant location (e.g. DBS, cochlear implant)
* Use of onabotulinum toxin A injections for the treatment of migraine in the past 3 months.
* Use of steroid infiltrations or IV administration in the past 3 months.
* Not pregnant, nursing or not using contraception

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation | 12 weeks
  The incidence of serious procedure, device and/or stimulation-related adverse events.
Effectiveness Evaluation | 12 weeks
  Difference between randomization arms, in proportion of subjects with ≥ 30% reduction in the number of Monthly Migraine Days (MMD).

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (2):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Resolve Pain, Buderim, Queensland
- Belgium (4):
  - Jessa Hasselt, Hasselt, Limburg
  - AZ Sint Jan Brugge, Bruges, West Vlaanderen
  - AZ Delta, Roeselare
  - ZAS Antwerpen, Campus Sint-Augustinus, Wilrijk
- Netherlands (2):
  - St. Antonius Nieuwegein, Nieuwegein
  - Erasmus MC Rotterdam, Rotterdam